CLINICAL TRIAL: NCT03421093
Title: A Multi-centre Real-world Non-interventional Observational Study to Evaluate Clinical Characteristics of the Chinese Patients With Lung Malignant Tumors Who Received Surgeries or Surgeries Plus Adjuvant Therapies
Brief Title: A Study to Evaluate Clinical Characteristics of Lung Cancer in Patients With Surgeries and Adjuvant Therapies
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Lunxu Liu, Professor, West China Hospital
Other Study IDs: TSCI-4
Record Dates: First submitted 2017-12-29; First posted 2018-02-05 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Chinese; surgeries; adjuvant therapies
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeries and adjuvant therapies: Surgeries or surgeries plus adjuvant therapies
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Surgeries or surgeries plus adjuvant therapies
  Other Names: Adjuvant therapies

SUMMARY:
The study was designed to evaluate effectiveness of the surgeries and adjuvant therapies after surgeries in the patients with lung malignant tumors

DETAILED DESCRIPTION:
The trial is a multi-centre real-world non-interventional observational study to evaluate effectiveness of the surgeries and adjuvant therapies after surgeries in the patients with lung malignant tumors via a retrospectively review method on the study data on patient demographic/tumor biological characteristics and clinical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old;
* Pathologically diagnosed lung malignant tumors after surgeries;
* Patients with lung surgeries;
* Patients with complete medical health records and follow-up visit information (at least one follow-up visit);

Exclusion Criteria:

* Patients who were not performed with surgeries;
* Pathologically diagnosed patients with benign diseases after surgeries;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung malignant tumors who were performed with surgeries
Sampling Method: Non-Probability Sample
Enrollment: 21777 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics of the patients with lung malignant tumors who received surgeries | 2014 - 2017
  Demographic characteristics of the patients with lung malignant tumors who received surgeries of thoracotomy, video-assistant thoracic surgery or robotic thoracic surgery as measured by:
  * Age
  * Gender
  * Payment types
  * Insurance types
  * Smoking history
  * Complications and symptoms of complications
  * Respiratory functions
  * Type of diagnoses

SECONDARY OUTCOMES:
Location of tumors and tumor sizes | 2014 - 2017
  Location of tumors and tumor sizes
Tumor clinical/pathological staging | 2014 - 2017
  Tumor clinical/pathological staging
Type of biomarkers | 2014 - 2017
  Type of biomarkers

OTHER OUTCOMES:
Differences in overall survivals of the patients with surgeries | 2014 - 2017
  Differences in perioperative overall survivals and overall survivals of the patients who received surgeries of thoracotomy, video-assistant thoracic surgery or robotic thoracic surgery
Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by tumor clinical/pathological staging | 2014 - 2017
  Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by tumor clinical/pathological staging
Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by location of tumors and tumor sizes | 2014 - 2017
  Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by location of tumors and tumor sizes
Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by duration and modes of surgeries | 2014 - 2017
  Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by duration and modes of surgeries
Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by type of insurances | 2014 - 2017
  Impact factors of patient survival in patients with tumor size =<2 cm who received surgeries as measured by type of insurances
Overall survival in the patients with tumor size =< 2cm who received surgeries | 2014 - 2017
  Overall survival in the patients with tumor size =< 2cm who received surgeries
Impact factors of patient survivals in the patients with N2 lung cancer with surgeries or surgeries plus adjuvant therapies | 2014 - 2017
  Impact factors of patient survivals in the patients with N2 lung cancer who received surgeries or surgeries plus adjuvant therapies
Overall survival in the patients with N2 lung cancer with surgeries or surgeries plus adjuvant therapies | 2014 - 2017
  Overall survival in the patients with N2 lung cancer who received surgeries or surgeries plus adjuvant therapies
Impact factors of patient survivals in the patients with small lung cancer with surgeries or surgeries plus adjuvant therapies | 2014 - 2017
  Impact factors of patient survivals in the patients with small lung cancer who received surgeries or surgeries plus adjuvant therapies
Overall survival in the patients with small lung cancer with surgeries or surgeries plus adjuvant therapies | 2014 - 2017
  Overall survival in the patients with small lung cancer who received surgeries or surgeries plus adjuvant therapies
Demographic characteristics of the patients with non-small cell lung cancer who were treated with chemotherapies, tyrosine kinase inhibitors, and other adjuvant therapies or were not treated with adjuvant therapies | 2014 - 2017
  Demographic characteristics of the patients with non-small cell lung cancer who were treated with chemotherapies, tyrosine kinase inhibitors, and other adjuvant therapies or were not treated with adjuvant therapies as measured by:
  * Age
  * Gender
  * Payment types
  * Insurance types
  * Smoking history
  * Complications and symptoms of complications
  * Respiratory functions
  * Type of diagnoses
Tumor clinical/pathological types | 2014 - 2017
  Tumor clinical/pathological types
Type of EGFR | 2014 - 2017
  Type of EGFR
ECOG scores | 2014 - 2017
  ECOG scores
1-year and 3-year overall survivals | 2014 - 2017
  1-year and 3-year overall survivals

CONTACTS AND LOCATIONS:
Overall Officials: Lunxun Liu, PhD, Principal Investigator — West China Hospital
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huaxi Technology University, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided